CLINICAL TRIAL: NCT05452564
Title: Phase II Study to Evaluate the Efficacy and Safety of Baricitinib for Reduction of HIV in the Central Nervous System
Brief Title: Baricitinib for Reduction of HIV - CNS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: William Tyor (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, William Tyor, Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004498; 1R01MH128158 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: Central Nervous System; Cerebrospinal Fluid; Baricitinib
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — baricitinib; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Potential participants will be pre-screened through review of the electronic medical record from Emory or Grady. Or if a potential participant receives care elsewhere, a release of medical information form will be signed and sent to the medical center that the individual goes to. The study team will enroll individuals who have well controlled HIV. Participants will then be randomized to either baricitinib or placebo.
  Patients randomized to Baricitinib group will receive Baricitinib at dose of 2 mg oral for ten weeks. Follow up visits will happen for both groups at weeks 1, 2, 4 and 10.
  Interventions: Drug: Baricitinib 2 MG Oral Tablet
- Placebo (Placebo Comparator): Potential participants will be pre-screened through review of the electronic medical record from Emory or Grady. Or if a potential participant receives care elsewhere, a release of medical information form will be signed and sent to the medical center that the individual goes to. The study team will enroll individuals who have well controlled HIV. Participants will then be randomized to either baricitinib or placebo.
  Patients randomized to the placebo group will receive 2 mg oral daily placebo for ten weeks. Follow up visits will happen for both groups at weeks 1, 2, 4 and 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib 2 MG Oral Tablet — Baricitinib, a Janus Kinase inhibitor drug for viral infections, will be administered orally to subjects randomized to this intervention. The dose will be 2 mg orally for ten weeks. This will be compared with placebo intervention. Follow up visits will take place at week 1,2,4 and 10.
  Other Names: Baricitinib
  Arms: Baricitinib
Drug: Placebo — Patients randomized to the placebo group will receive 2 mg oral daily placebo for ten weeks. Follow up visits will happen for both groups at weeks 1, 2, 4 and 10.
  Arms: Placebo

SUMMARY:
There is still no cure for the human immunodeficiency virus (HIV). While combination antiretroviral therapy (cART) is effective in decreasing deaths from HIV, infected individuals face a lifetime of treatment and many potential complications including end organ diseases such as HIV-associated neurocognitive disorders. HIV infection is controllable with antiretroviral therapy (ART), but ART cannot eliminate HIV reservoirs. Thus, there is no available cure for HIV. There is a large and growing body of evidence that the central nervous system (CNS) is an HIV reservoir site and a barrier to HIV eradication. Our group has done extensive pre-clinical work with janus-kinase (JAK 1/2) inhibitors. This includes baricitinib, which is an orally available, FDA-approved drug for rheumatoid arthritis. Evidence suggests that this drug has activity against HIV in the central nervous system (CNS). In our recently completed pilot study, we showed that baricitinib crosses the blood brain barrier (BBB) and decreases HIV CNS persistence in the brain.

Using bloodwork, neurocognitive testing, MRIs and lumbar punctures, we plan to evaluate the change in central nervous system HIV after treatment with baricitinib versus placebo. We will also evaluate changes in neuroimaging, inflammation in blood and cerebrospinal fluid (CSF), and neuropsychological performance after treatment with baricitinib versus placebo.

Evidence shows that the central nervous system is one of the reservoir sites that enables the HIV virus to persist in the body even after years of treatment. In order to attack this reservoir and eventually find a cure, it is vital to learn if certain medications can suppress HIV in the CNS.

DETAILED DESCRIPTION:
HIV infection is controllable with antiretroviral therapy (ART), but ART cannot eliminate HIV reservoirs. Thus, there is no available cure for HIV. There is a large and growing body of evidence that the central nervous system (CNS) is an HIV reservoir site and a barrier to HIV eradication. HIV DNA is commonly found in brain from people with HIV (PWH) on suppressive ART. HIV genetic compartmentalization occurs in both the brain and CSF, showing that CNS HIV is distinct from peripheral sources such as blood. Multiple studies have demonstrated that CSF HIV RNA can be detected at very low levels during suppressive ART. A study from the AIDS Clinical Trials Group (ACTG) found HIV DNA in CSF cells from approximately 50% of PWH on suppressive ART, a finding that was associated with neurocognitive impairment. The study team's group recently demonstrated a significant advance in quantitating HIV from the CSF. Specifically, CSF cell associated HIV RNA was quantifiable in 90% and CSF HIV DNA was quantifiable in 80% of PWH on suppressive ART. Based on these multiple lines of evidence that the CNS is an HIV reservoir, more research is needed on therapies that have the potential to target the CNS reservoir.

The study team has performed extensive pre-clinical and clinical work on the Janus Kinase (Jak 1/2) inhibitor drug class for viral infections. This includes work on ruxolitinib and baricitinib, two FDA approved orally bioavailable agents for myelofibrosis and polycythemia vera (ruxolitinib) as well as rheumatoid arthritis (baricitinib). The investigators have evaluated their potential to target HIV in the CNS in vitro, ex vivo, and in vivo Specifically, the study team has demonstrated that these agents block HIV replication and infection in key CNS cells, reduce the lifespan of HIV CNS reservoirs, and block reservoir reseeding. In vivo, the study team has shown in the murine model that baricitinib decreases CNS HIV and reverses behavioral abnormalities associated with HIV, which correlates with reversal of phenotypic markers of brain inflammation. This has also demonstrated that baricitinib reaches therapeutic CNS concentrations in the rhesus macaque model (including in brain parenchyma) as well as in humans. In a recently published multi-site Phase 2a ACTG-sponsored study with ruxolitinib (A5336, n = 60),the research group demonstrated that ruxolitinib is safe, well-tolerated, and reduces key markers of immune activation. New data that ruxolitinib decreased the peripheral HIV reservoir in a subset of A5336 participants provides even more evidence for this drug class to be included in eradication strategies. However, A5336 did not have any CNS assessments. The investigators now propose to study baricitinib, one of the most promising Jak 1/2 inhibitors with once daily dosing, renal clearance, and a more favorable safety/ pharmacokinetic profile, as a therapy to decrease the HIV CNS reservoir in PWH with durable virologic suppression on ART.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected on continuous ART with plasma HIV RNA <200 copies/ml for at least 12 months (on at least two previous clinic visits and confirmed at screening). If a viral load is documented from a CLIA-certified laboratory 14 days before screening, then this result can be used in place of the screening lab result.
2. Current CD4+ > 350 cells/microliter for at least twelve months (on at least two previous clinic visits and confirmed at screening). If a CD4 count is documented from a CLIA-certified laboratory 30 days before screening, then this result can be used in place of the screening lab result.
3. Women of reproductive age will have a negative pregnancy test at study entry and agree to contraception while on the study drug. Women who are at least 50 years of age and who have been amenorrheic for at least 12 months will not be required to agree to contraception to participate.

Exclusion Criteria:

1. < 18 years of age or > 65 years of age
2. Pregnancy or breastfeeding
3. Significant hematological abnormalities at screening (ANC < 1500, Hgb<10, platelet< 100,000)
4. History of progressive multifocal leukoencephalopathy
5. Untreated latent tuberculosis infection (which will be screened for before entry). If there is a prior positive test, the test does not need to be repeated at screening.
6. Immunosuppressive medications (including corticosteroids) and anticoagulants (aspirin acceptable) within 1 month. A partial list is provided in the SOP for staff, but otherwise, if there is a question it will be adjudicated by the Investigator(s).
7. History of deep venous thrombosis
8. Cardiovascular disease:

   1. Coronary artery disease or history of myocardial infarction, no exclusion if greater than 3 months
   2. Congestive heart failure with left ventricular ejection fraction ≤40% per American Heart Association guidelines-- no exclusion if greater than 3 months
   3. Ever a history of stroke
9. Hematologic malignancies including lymphoma and leukemia which have no evidence of cure or are at least in remission for > 5 years
10. Major surgery within 8 weeks before screening or will require major surgery during the study
11. Current or recent (<4 weeks before randomization) clinically serious viral (including COVID-19), a bacterial, fungal, or parasitic infection or any other active or recent infection. History of untreated syphilis infection. If an RPR was negative in the 3 months before screening, then an RPR is not needed at screening
12. Symptomatic herpes simplex at the time of randomization
13. Symptomatic herpes zoster infection within 12 weeks before randomization.
14. History of disseminated/complicated herpes zoster (for example, ophthalmic zoster or CNS involvement).
15. Positive test for hepatitis B virus (HBV) defined as:

    1. positive for hepatitis B surface antigen (HBsAg), or
    2. positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA)
16. Hepatitis C virus (HCV) chronic infection (hepatitis C antibody-positive and HCV ribonucleic acid [RNA]-positive), ever.
17. Cirrhosis of the liver from any cause
18. Any of the following specific abnormalities on screening laboratory tests:

    1. ALT or AST >2 x upper limits of normal (ULN)
    2. alkaline phosphatase (ALP) ≥2 x ULN
    3. total bilirubin ≥1.5 x ULN (except patients on atazanavir, who must have total bilirubin <2 x ULN)
    4. International Normalized Ratio (INR) > 1.5
    5. Absolute Neutrophil Count (ANC) <1000 cells/mm3, confirmed on repeat testing.
19. Chronic kidney disease with eGFR <40 mL/min/1.73 m2 (note that the dose of baricitinib will be reduced to 1 mg daily in participants with GFR between 40 and 60). Specifically, the CKD-EPI without race-based equation is used
20. Current dependence on illicit drugs except for marijuana
21. Bleeding disorders such as Von Willebrand's Disease, hemophilia, or other coagulopathies as determined by history.
22. Any evidence of a mass lesion by history that could lead to increased intracranial pressure and evidence of trauma to the lumbar vertebra (see LP exclusion criteria above) by history. - no lumbar trauma or surgery in the last 60 days, but this will be adjudicated by Investigator(s) if need be.
23. Population: The study team will not include any of the following groups:

    * Adults unable to consent
    * Individuals who are not yet adults (infants, children, teenagers)
    * Pregnant women
    * Prisoners
    * Cognitively impaired or Individuals with Impaired Decision-Making Capacity
    * Individuals who are not able to clearly understand English
    * Community Participation (if applicable)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Changes in CSF integrated proviral DNA | Baseline and study week 10
  The study team will obtain up to 40 milliliters (ml) of CSF from individuals who weigh at least 60 kilograms, otherwise, they will draw up to 30 ml of CSF.
  CSF integrated proviral DNA (IPDA and Alu-PCR) will be assessed: Integrated proviral DNA will be performed using existing methods in the clinical research group, which employ the Alu-PCR real-time platform, with a limit of 3 copies. Integrated proviral DNA assay (IPDA) to measure the replication-competent reservoir will be used with digital droplet PCR methodology.

SECONDARY OUTCOMES:
Changes in CSF HIV RNA by single copy assay | Baseline and study week 10
  This method is based on a proprietary protocol which is used in conjunction with a commercial HIV-1 RNA easyQ reagent kit (bioMerieux Inc, Lyon, France). Briefly, a specimen of up to 2 ml of human plasma or CSF is added to lysis buffer containing guanidine thiocyanate. HIV-1 RNA is extracted in combination with the easyMAG platform (bioMerieux, Inc). Eluates containing HIV-1 RNA are aliquoted into 0.5 mL reaction tubes and amplified using 3 enzymes: T7 RNA polymerase, avian myeloblastosis virus reverse transcriptase, and RNase H. Molecular beacons targeting the pol/gag region of HIV-1 RNA are used for amplification and detection by isothermal reactions at 41oC. HIV-1 RNA level is quantified in conjunction with the NucliSENS easyQ HIV-1 v2.0 Director software and a proprietary algorithm developed by bioMONTR Labs. The dynamic range of this HIV-1 assay is 1-5,000,000 copies/mL of 0.73 - 1600 HIV-1 copies /μl. The HIV-1 copy number is normalized per one million of WBCs.
Changes in HIV tat protein in CSF | Baseline and study week 10
  The study team will obtain up to 40 milliliters (ml) of CSF from individuals who weigh at least 60 kilograms, otherwise we will draw up to 30 ml of CSF.
  HIV Tat in the CSF will be quantified according to published methods for ELISA to measure HIV Tat in human CSF.
Changes in CSF HIV cell-associated RNA by Double-R assay. | Baseline and study week 10
  The study team will obtain up to 40 milliliters (ml) of CSF from individuals who weigh at least 60 kilograms, otherwise, they will draw up to 30 ml of CSF.
  Briefly, after the isolation of Peripheral blood mononuclear cells (PBMC) and cells from CSF, samples will be resuspended in phosphate-buffered saline and stored for shipment in O-ring tubes. RNA will then be extracted using the Maxwell rapid sample concentrator (RSC) automated extraction platform. White Blood Cells (WBC) will be counted after red blood cell lysis using TC20 Automated Cell Counter, and these counts will be used to normalize the HIV-1 RNA results as copy numbers/106 cells. HIV-1 copy number per patient sample, in duplicate, is determined from a standard curve generated with HIV-1 plasmid controls, with a range of 0.73 - 1600 HIV-1 copies /μl. The HIV-1 copy number is normalized per one million of WBCs.
Changes in CSF HIV cell associated CSF HIV DNA by Double-R assay. | Baseline and study week 10
  The study team will obtain up to 40 milliliters (ml) of CSF from individuals who weigh at least 60 kilograms, otherwise they will draw up to 30 ml of CSF.
  Briefly, after the isolation of Peripheral blood mononuclear cells (PBMC) and cells from CSF, samples will be resuspended in phosphate-buffered saline and stored for shipment in O-ring tubes. DNA will then be extracted using the Maxwell rapid sample concentrator (RSC) automated extraction platform. WBCs will be counted after red blood cell lysis using TC20 Automated Cell Counter, and these counts will be used to normalize the HIV-1 DNA results as copy numbers/106 cells. HIV-1 copy number per patient sample, in duplicate, is determined from a standard curve generated with HIV-1 plasmid controls, with a range of 0.73 - 1600 HIV-1 copies /μl. The HIV-1 copy number is normalized per one million of WBCs.
Changes in CSF cell associated DNA | Baseline and study week 10
  The study team will obtain up to 40 milliliters (ml) of CSF from individuals who weigh at least 60 kilograms, otherwise we will draw up to 30 ml of CSF.
  Cell associated DNA will be performed according to standard existing protocols using real-time PCR with a limit of detection of five copies.
Changes in Blood HIV cell associated RNA by Double-R assay | Baseline and study week 10
  Changes in the blood between baseline and week ten after study medication. Briefly, after isolation of Peripheral blood mononuclear cells (PBMC) and cells from patient's blood sample, samples will be resuspended in phosphate buffered saline and stored for shipment in O-ring tubes. RNA will then be extracted using the Maxwell rapid sample concentrator (RSC) automated extraction platform. WBCs will be counted after red blood cell lysis using TC20 Automated Cell Counter, and these counts will be used to normalize the HIV-1 RNA results as copy numbers/106 cells. HIV-1 copy number per patient sample, in duplicate, is determined from a standard curve generated with HIV-1 plasmid controls, with a range of 0.73 - 1600 HIV-1 copies /μl. The HIV-1 copy number is normalized per one million of WBCs.
Changes in Blood HIV cell associated DNA by Double-R assay | Baseline and study week 10
  Changes in the blood between baseline and week ten after study medication. Briefly, after isolation of Peripheral blood mononuclear cells (PBMC) and cells from the patient's blood sample, samples will be resuspended in phosphate buffered saline and stored for shipment in O-ring tubes. DNA will then be extracted using the Maxwell rapid sample concentrator (RSC) automated extraction platform. WBCs will be counted after red blood cell lysis using TC20 Automated Cell Counter, and these counts will be used to normalize the HIV-1 DNA results as copy numbers/106 cells. HIV-1 copy number per patient sample, in duplicate, is determined from a standard curve generated with HIV-1 plasmid controls, with a range of 0.73 - 1600 HIV-1 copies /μl. The HIV-1 copy number is normalized per one million of WBCs.
Changes in Blood cell associated DNA | Baseline and study week 10
  Change in the blood between baseline and week ten after study medication. Cell associated DNA will be performed according to standard existing protocols using real-time PCR with a limit of detection of five copies.
Change in HIV DNA levels by Integrated proviral DNA assay | Baseline and study week 10
  Change in the blood between baseline and week ten after study medication. The study team will obtain up to 40 milliliters (ml) of CSF from individuals who weigh at least 60 kilograms, otherwise we will draw up to 30 ml of CSF.
  Blood integrated proviral DNA (IPDA and Alu-PCR) will be assessed: Integrated proviral DNA will be performed using existing methods in our group, which employ the Alu-PCR real-time platform, with a limit of 3 copies. Integrated proviral DNA assay (IPDA) to measure the replication competent reservoir will be used with digital droplet PCR methodology
Changes in Blood HIV RNA by single copy assay | Baseline and study week 10
  This method is based on a proprietary protocol which is used in conjunction with a commercial HIV-1 RNA easyQ reagent kit (bioMerieux Inc, Lyon, France). Briefly, a specimen of up to 2 ml of human plasma or CSF is added to lysis buffer containing guanidine thiocyanate. HIV-1 RNA is extracted in combination with the easyMAG platform (bioMerieux, Inc). Eluates containing HIV-1 RNA are aliquoted into 0.5 mL reaction tubes and amplified using 3 enzymes: T7 RNA polymerase, avian myeloblastosis virus reverse transcriptase, and RNase H. Molecular beacons targeting the pol/gag region of HIV-1 RNA are used for amplification and detection by isothermal reactions at 41oC. HIV-1 RNA level is quantified in conjunction with the NucliSENS easyQ HIV-1 v2.0 Director software and a proprietary algorithm developed by bioMONTR Labs. The dynamic range of this HIV-1 assay is 1-5,000,000 copies/mLof 0.73
Changes in Blood indirect viral markers: anti-HIV antibody levels | Baseline and study week 10
  Change in HIV and inflammation levels in the blood between baseline and week ten after study medication.
  Blood HIV antibodies by LIPS assay (gp120, integrase, protease, and p24) will be assayed. The LIPS assay uses recombinant chimeric fusion proteins with luciferase producing light and specific antigens for quantitative detection of antibodies.
Changes in Blood indirect viral markers: HIV specific T cells | Baseline and study week 10
  Change in HIV and inflammation levels in the blood between baseline and week ten after study medication Fresh Human peripheral blood mononuclear cells (PBMC) will be cultured in the presence or absence of overlapping peptides which induces broad, non-specific T-cell activation. In addition to cytokine production (focusing on TNFα, IFNγ, and IL-6 measured with Quanterix technology). Researchers will measure cell surface markers by flow cytometry.
Changes in Blood CXCL10 | Baseline and study week 10
  Change in levels in the blood between baseline and week ten after study medication.
  The study team will measure CXCL10 from participants blood samples, in the setting of HIV using single molecule array technology by Quanterix.
Changes in Blood Neopterin | Baseline and study week 10
  Change in levels in the blood between baseline and week ten after study medication.
  The study team will measure neopterin in the setting of HIV using the enzyme linked immunosorbent assays produced by Uman diagnostics, R&D Systems (ultra-sensitive), and Themo Fisher.
Changes in Blood IL-7 | Baseline and study week 10
  Change in levels in the blood between baseline and week ten after study medication.
  This will be measured using mesoscale discovery platform.
Changes in Blood IL-15 | Baseline and study week 10
  Change in levels in the blood between baseline and week ten after study medication.
  This will be measured using mesoscale discovery platform.
Changes in Stroop Test (Color Naming and Color-Word) | Baseline and study week 10
  In psychology, the Stroop effect is the delay in reaction time between congruent and incongruent stimuli.
  The effect has been used to create a psychological test (the Stroop test) that is widely used in clinical practice and investigation.
  A basic task that demonstrates this effect occurs when there is a mismatch between the name of a color (e.g., "blue", "green", or "red") and the color it is printed on (i.e., the word "red" printed in blue ink instead of red ink). When asked to name the color of the word it takes longer and is more prone to errors when the color of the ink does not match the name of the color.
  Word, color, and color-word T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal." In order for one score to be considered "higher" or "lower" than another, a 10 point or greater T score difference is required.
Changes in Hopkins Verbal Learning Test II (Learning and Recall) | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided.
  The Hopkins Verbal Learning Test-Revised (HVLT-R) is used to assess acquisition and delayed recall. The HVLT-R is a list learning test, which consists of 12 nouns within three semantic groups. The acquisition variable consists of three acquisition trials in which the administrator reads the words aloud and then asks the child to repeat as many as he/she can remember in any order. A delayed recall trial is introduced after 20-25 min, in which the child is asked to simply retrieve as many of the words listed in the acquisition trial as he/she can remember. The children are not informed about the delayed recall trial beforehand. Lower raw scores indicate difficulties with the task.
Changes in Brief Visuospatial Test (Learning and Recall) | Baseline and study week 10
  The Brief Visuospatial Memory Test (BVMT) is a commonly used assessment tool to measure visuospatial learning and memory abilities.
  In three Learning Trials, the respondent views the stimulus page for 10 seconds and is asked to draw as many of the figures as possible in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Last, a Recognition Trial, in which the respondent is asked to identify which of 12 figures were included among the original geometric figures, is administered.
  An optional Copy Trial may be administered to screen for severe visuoconstructive deficits and to help in scoring recall responses.
  12 scores may be derived from BVMT-R performance. Recall performance is recorded for each of the immediate recall trials (Trial 1, Trail 2, and Trial 3) and for the delayed recall trial (Delayed Recall).
  The recall scores are combined to form three additional summary measures of learning and memory.
Changes in Trailmaking | Baseline and study week 10
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It requires a subject to connect a sequence of 25 consecutive targets on a sheet of paper or computer screen. There are 2 parts to the test: in the first, the targets are all numbers from 1 to 25 and the test taker needs to connect them in sequential order; in the second part, the dots go from 1 to 13 and include letters from A to L. As in the first part, the patient must connect the dots in order while alternating letters and numbers, as in 1-A-2-B-3-C..., in the shortest time possible without lifting the pen from the paper. If the subject makes an error, the administrator corrects them before moving on to the next dot.
  The subject's goal is to finish both parts as quickly as possible, with the time taken to complete the test being used as the primary performance metric. Scoring is based on time taken to complete the test (e.g. 35 seconds yielding a score of 35) with lower scores being better
Changes in Digit Symbol Test | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided.
  The Digit Symbol Substitution Test (DSST) is a paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located on the top of the page. The subject copies the symbol into spaces below a row of numbers. The number of correct symbols within the allowed time, usually 90 to 120 seconds, constitutes the score.
Changes in Letter Number Sequencing Test | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided.
  Letter-number sequencing is a subtest of the WAIS (Wechsler Adult Intelligence Scale) and the WISC (Wechsler Intelligence Scale for Children). It is a test that measures an individual's short-term memory skills in being able to process and re-sequence information. The task involves hearing a series of letters and digits, and then reporting back the stimuli with the letters in alphabetical order, and digits in ascending numerical order. The task is traditionally administered orally, but recent studies have administered versions of the tasks visually by displaying stimuli on a computer screen. Results suggest that performance differences on the Letter-Number Sequencing task may arise as a function of language background and task administration modality
Changes in Wisconsin Card Sorting Test | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided.
Changes in Grooved Pegboard Test | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided.
  The Grooved Pegboard Test (GPT) is used primarily as a measure of motor functioning, but some research indicates that performance on this test my also reflect cognitive factors, particularly attention and executive functioning.
  This manipulative dexterity test contains twenty-five holes with randomly positioned slots and pegs which have a key along one side. Pegs must be rotated to match the hole before they can be inserted.
  This procedure measures performance speed in a fine motor task by examining both sides of the body, inferences may be drawn regarding possible lateral brain damage.
  The test requires more complete visual motor coordination than most of our pegboards and has been used in several neuropsychological test batteries, in student labs, and as a screening technique in industrial environment.
Changes in Letter and category fluency test | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided.
Changes in Beck Depression Inventory II (BDI-II) | Baseline and study week 10
  This will be performed in a quiet exam room. Participants will have the opportunity to take breaks as needed and snacks will be provided. The BDI-II is a widely used 21-item self-report inventory measuring the severity of depression in adolescents and adults.
  The questionnaire consists of 21 questions with answers ranging from 0 to 3. Scores are later analyzed by adding all scores and comparing to ranges :
  0-10:These ups and downs are considered normal 11-16:Mild mood disturbance 17-20:Borderline clinical depression 21-30:Moderate depression 31-40: Severe depression over 4: Extreme depression
Changes in MRI neuroimaging findings | Baseline and study week 10
  Brain structure and function will be evaluated using magnetic resonance (MR) data acquired on a 7T Siemens Terra scanner with a multi-channel head coil. Data acquisition will include sequences for structural imaging, resting state functional MRI, diffusion imaging, perfusion imaging, and magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: William Tyor, MD, Principal Investigator — Professor
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Medical and social history, laboratory results, imaging results, neuropsychological test results
Supporting Information: Study Protocol, SAP
Time Frame: At the end of the study until 2027
Access Criteria: Qualified investigators for secondary analyses not related to the primary aims of the study following Emory University guidelines